CLINICAL TRIAL: NCT07037355
Title: Association Between Hand-Eye Coordination and Handgrip Strength in Children Post-Healing of Distal Radius Greenstick Fractures: A Cross-Sectional Study
Brief Title: Association Between Hand-Eye Coordination and Handgrip Strength in Children Post-Healing of DRGF
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: DPT/Batch-Fall20/1014
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Radius Fractures
MeSH Terms: conditions — Radius Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Handgrip Strength and Hand-Eye Coordination Assessment
  Interventions: Combination Product: Handgrip Strength and Hand-Eye Coordination Assessment

INTERVENTIONS:
Combination Product: Handgrip Strength and Hand-Eye Coordination Assessment — Children underwent standardized testing to assess functional recovery post-healing of distal radius greenstick fractures.

SUMMARY:
The study investigates whether hand-eye coordination is related to handgrip strength in children (aged 5-12 years) after they have healed from distal radius greenstick fractures. This is important because both strength and coordination are crucial for a child's full functional recovery after such fractures.

Cross-sectional analytical study Orthopedic and physiotherapy departments in Lahore 84 children (convenience sampling)

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-12 years
* Radiologically confirmed healed distal radius greenstick fractures
* Ability to perform handgrip and hand-eye coordination tests
* Parental consent and child assent

Exclusion Criteria:

* Acute pain or swelling at the time of testing
* Current medications affecting bone/muscle function
* Neuromuscular or developmental disorders
* History of previous upper limb fractures or surgeries

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Handgrip Strength and Hand-Eye Coordination Assessment in the Association Between Hand-Eye Coordination and Handgrip Strength in Children Post-Healing of Distal Radius Greenstick Fractures: A Cross-Sectional Study
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Beery-Buktenica Developmental Test of Visual-Motor Integration | 6 Month
  (Beery VMI): Provides standard scores and percentile ranks:
  129: Very High (2% of age group)
  120-129: High (7%)
  110-119: Above Average (16%)
  90-109: Average (50%)
  80-89: Below Average (16%)
  70-79: Low (7%)
  <70: Very Low (2%)

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University CRC, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No